CLINICAL TRIAL: NCT02198105
Title: Registry of Cutting Balloon and DCB Intervention in Femoropopliteal Stenosis/Occlusion.
Acronym: DEBTRAK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Caritasklinik St. Theresia (Other)
Responsible Party: Principal Investigator, Magnus Baumhäkel, PD Dr. med. Magnus Baumhäkel, Caritasklinik St. Theresia
Other Study IDs: DEBTRAK-Registry
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Peripheral Artery Disease; Femoropoliteal Stenosis/Occlusion; Cutting-balloon; Drug-coated-balloon
Keywords: PAD; femoropoliteal stenosis/occlusion; cutting-balloon; drug-coated-balloon
MeSH Terms: conditions — Peripheral Arterial Disease; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Femoropopliteal stenosis: Consecutive patients with symptomatic peripheral artery disease due to femoro-popliteal stenosis/occlusion.
  Intervention with Cutting-Balloon-PTA (VascuTrak) and Drug Coated Ballon-PTA.
  Interventions: Device: Cutting-Balloon-PTA (VascuTrak) and Drug Coated Ballon PTA

INTERVENTIONS:
Device: Cutting-Balloon-PTA (VascuTrak) and Drug Coated Ballon PTA — Interventional procedure:
  1. PTA with Cutting-Balloon (60-120 seconds).
  2. PTA with DC-Balloon (60 seconds).
  Technical success is defined as
  1. no recoil >30%
  2. no dissection >Type B
  3. no stenting >30% of lesion length.

SUMMARY:
Observational registry including patients with peripheral artery disease due to femoro-popliteal stenosis or occlusion treated with cutting ballon- and subsequent drug-coated-ballon-percutaneous-transluminal-angioplasty (PTA).

DETAILED DESCRIPTION:
The registry includes consecutive patients with symptomatic peripheral artery disease due to femoro-popliteal stenosis or occlusion treated with cutting ballon- and subsequent drug-coated-ballon-percutaneous-transluminal-angioplasty (PTA).

Interventional procedure:

1. PTA with Cutting-Balloon (60-120 seconds).
2. PTA with Drug-Coated-Balloon (60 seconds).

Technical success is defined as

1. no recoil >30%
2. no dissection >Type B
3. no stenting >30% of lesion length.

Follow-up of patients after 6 months and 12 months (ABI, Rutherford-classification, MACE, TLR, TVR, Binary Restenosis).

ELIGIBILITY:
Inclusion Criteria:

* peripheral artery disease (PAD) with femoro-popliteal stenosis >70% or occlusion (vessel diameter 4-6mm)
* age 18-99
* informed consent

Exclusion Criteria:

* proximal / iliacal stenosis
* stenosis/occlusion of all arteries below the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic peripheral artery disease due to femoro-popliteal stenosis or occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Clinically driven target lesion revascularization (TLR) | 6 months
  clinically driven target lesion revascularization

SECONDARY OUTCOMES:
clinically driven target vessel revascularization (TVR) | 6 months
  TVR
Binary restenosis | 6 months
  Peak Systolic velocity (PSV) >2.4
Change in Ankle Brachial Index (ABI) | 6 months
  Change in ankle brachial index from baseline.
Change in Rutherford-classification | 6 months
  Change in Rutherford-Classification from Baseline (I-VI)
major cardiac adverse events | 6 months
  myocardial infarction, stroke, death, cardiovascular death
Amputation | 6 months
clinically driven target vessel revascularization (TVR) | 12 months
Clinically driven target lesion revascularization (TLR) | 12 months
Binary restenosis | 12 months
Change in Ankle Brachial Index (ABI) | 12 months
Change in Rutherford-classification | 12 months
major cardiac adverse events | 12 months
  myocardial infarction, stroke, death, cardiovascular death
Amputation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Baumhäkel, MD, Principal Investigator — CaritasKlinikum, St. Theresia Saarbrücken, Germany
Locations (1):
- CaritasKlinikum, St. Theresia, Saarbrücken, Saarland, Germany